CLINICAL TRIAL: NCT05979974
Title: Efficacy of High Energy Density Pulse Electromagnetic Field for Patients With Frozen Shoulder: A Double-blinded, Randomized Controlled Trail
Brief Title: High Energy Density Pulse Electromagnetic Field for Patients With Frozen Shoulder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find participants willing to join the trial.
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Director, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A202305106
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; high energy density pulse electromagnetic field
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy and high-PEMF (Experimental): The patient undergoes physiotherapy and high-PEMF therapy twice a week, for a duration of three weeks.
  Interventions: Device: High energy density pulse electromagnetic field; Other: physiotherapy
- physiotherapy and sham high-PEMF (Sham Comparator): The patient undergoes physiotherapy and sham high-PEMF therapy twice a week, for a duration of three weeks.
  Interventions: Other: physiotherapy; Device: sham High energy density pulse electromagnetic field

INTERVENTIONS:
Device: High energy density pulse electromagnetic field — The treatment coil is placed over the shoulder region at the maximum pain point for 9 minutes. A high energy of high-PEMF with a rate of 3 pulse per second is applied to the patient.
  Arms: physiotherapy and high-PEMF
Other: physiotherapy — Physiotherapy such as shoulder passive and active-assisted range of motion (ROM) exercises, Pendulum exercises, Codman's exercises and Cross-body reach exercises. Under the physiotherapist's guidance, the patient receives the training session about 30 minutes every time.
Device: sham High energy density pulse electromagnetic field — The sham treatment coil is placed over the shoulder region at the maximum pain point for 9 minutes. The setting is the same as the experimental group(high energy, a rate of 3 pulse per second) with the difference that the energy output doesn't export to the patient.
  Arms: physiotherapy and sham high-PEMF

SUMMARY:
The aim of our study is to investigate the efficacy of high energy density pulse electromagnetic field for patients with frozen shoulder

DETAILED DESCRIPTION:
Frozen shoulder causes shoulder pain and limited range of motion(ROM). It is thought to afflict between 2 and 5% of the general population. Individuals of middle age are most often affected, typically during the 5th to 7th decades of life. Typical symptoms include gradual onset of shoulder pain, limited shoulder ROM at least in two or more directions (especially in external rotation). In the case of primary adhesive capsulitis, the disease is usually self-limiting, and typically lasts 18-24 months. However, persistent symptoms and movement restriction beyond 3 years have been reported in up to 40% of patients, with up to 15% of patients suffering permanent disability. Therefore, an effective treatment is necessary to treat the shoulder pain and disability caused by frozen shoulder. High energy density pulse electromagnetic field (High-PEMF), different from traditional PEMF, includes characteristics as following:

1. The short pulse duration (50μs) with a damped oscillation
2. The broad bandwidth(200kHz~300MHz) with a basic frequency 240kHz
3. High voltages (up to 40 kV) and peak currents (up to 10 kA) arise in the applicator spool
4. Delivery of energy per pulse of about 96Ws (Joule) with a magnetic flux density of 50~100mT
5. Depth penetration for tissue and organ up to 20 cm

It has been applied in chronic tendinopathy with positive outcomes. However, few studies support its application in the setting of frozen shoulder. Hence, the aim of our study is to investigate the efficacy and the underlying possible mechanism of High-PEMF for patients with frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Frozen shoulder is diagnosed by physicians based on the patient's medical history, physical examination, X-ray, and ultrasound reports.
2. The symptoms persist for more than 3 months.
3. There is a reduction of at least 30 degrees in at least two of the affected shoulder joint angles compared to the angles of the healthy side: shoulder flexion, abduction, and external rotation.

Exclusion Criteria:

1. Shoulder musculoskeletal ultrasound reveals a full-thickness tear or massive tear of the shoulder rotator cuff tendons or calcific tendinitis.
2. Systemic rheumatic disease.
3. History of shoulder fracture or previous surgical treatment of the shoulder joint.
4. Acute cervical nerve root compression.
5. Patients with instability (e.g., those with symptoms of internal bleeding) or cancer patients.
6. Received shoulder injections for treatment within the past 3 months.
7. Impaired cognitive function that prevents the patient from providing informed consent or participating in rehabilitation therapy.
8. Pregnant or breastfeeding women.
9. Meets any of the contraindications for high-energy electromagnetic pulse therapy: organ transplant recipients; individuals with implanted cardiac pacemakers, defibrillators, metal implants (such as stents), cochlear implants, and insulin supplementation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in pain Visual Analogue Scale(VAS) | the change from baseline, post-intervention immediately, post-intervention 1, 3, 6 months
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. "0" means painless and "10" means extremely painful.

SECONDARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | the change from baseline, post-intervention immediately, post-intervention 1, 3, 6 months
  Shoulder function and disability were evaluated using the Chinese version of the Shoulder Pain and Disability Index (SPADI), a self-report questionnaire that yields pain and disability domain and total scores. The SPADI includes five questions on pain and eight questions on disability, referring to various problems with the shoulder encountered over the preceding week. Each item's score ranges from 0 (no pain/normal) to 10 (maximal pain/disability), with total scores of pain from 0-50 and disability from to 0-80. A higher score shows more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Liang cheng Chiang, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General
Locations (1):
- Tri-service general hospital, Taipei, Taiwan